CLINICAL TRIAL: NCT00382044
Title: Audit of the Effect of Changing From IV to SC Administration of Erythropoiesis Stimulating Agents in Haemodialysis Patients - Real Life Clinical Experience
Brief Title: Audit of the Effect of Changing From IV to SC Administration of ESA's in Haemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Sir Charles Gairdner Hospital (Other)
Responsible Party: Dr Neil Boudville, Sir Charles Gairdner Hospital
Other Study IDs: NB-06-10
Record Dates: First submitted 2006-09-27; First posted 2006-09-28 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Kidney Failure, Chronic; Anemia
Keywords: Kidney Failure, Chronic; Dialysis; Anemia; epoetin
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia | interventions — Epoetin Alfa; epoetin beta; Darbepoetin alfa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Eprex; Neorecormon; Aranesp

SUMMARY:
The purpose of this study is to audit the effects of changing all hemodialysis patients from intravenous to subcutaneous administration of ESA's, to ensure that a cost-saving is achieved and that this does not occur at the expense of anemia control. The dose changes will occur according to usual clinical care of patients and not along a protocol.

DETAILED DESCRIPTION:
Background

Erythropoietin Stimulating Agents (ESAs) are widely used by chronic kidney disease patients who suffer with renal associated anemia. Until recently there have been only two ESAs currently available in the Australia: epoetin alfa/Eprex® (Janssen Cilag) and darbepoetin alfa/Aranesp® (Amgen). Following expiry of the Eprex® patent earlier this year another agent, epoetin beta/NeoRecormon® (Roche) has also become available . While ESAs provides significant benefits to the patients, with reduced morbidity and mortality, it comes at a considerable economic cost.

Clinical evidence indicates that the SC route of epoetin (epoetin alfa and epoetin beta) is more efficient clinically than IV, which is reflected by smaller epoetin dose requirements (e.g. Kaufman et al 1998; NeoRecormon Product Information dated 6 December 2005). Whilst the dose reduction for patients changing from IV to SC epoetin is variable, a recent meta-analysis showed 30% dose reduction by the SC route, resulting in significant cost savings (Besarab et al 2002). Furthermore, the NeoRecormon Product Information states that 'generally the subcutaneous maintenance dose is approximately 20% to 35% lower than the intravenous maintenance dose'. However, studies monitoring the conversion patients treated with SC epoetin alfa to IV epoetin alfa showed only 15% increase in dose requirements in Swedish haemodialysis patients (Torbjörn et al 2005) and 8.7% in Australian hemodialysis patients (Pussell and Walker 2003). Unlike epoetin, there is no difference in efficiency of darbepoetin alfa by route of administration (Vanrentergham et al 2002; Cervelli et al 2005).

Prior to 2002, ESAs were primarily administered by the subcutaneous route of administration, due to lower dose requirements and thus cost savings for epoetin alfa. However, in 2002 the subcutaneous route of epoetin alfa in chronic kidney disease was contraindicated due to an increase in the incidence of cases of anti-Epo antibody medicated pure red cell aplasia (PRCA) associated with subcutaneous use of the product between 1998 and 2002. Since then the majority of hemodialysis patients in Australia have been treated with ESAs by the intravenous route of administration. Recently the manufacturers identified the probable cause of increased immunogenicity of epoetin alfa and corrected for it (Boven et al 2005). Consequently, the TGA reinstated the use of subcutaneous epoetin alfa in chronic kidney disease patients in mid-2005 (240th ADEC Meeting Recommendations, June 2005). By converting hemodialysis patients back to subcutaneous ESA administration this may lead to considerable cost-savings: for every 100 patients on 11,200IU epoetin a week (current Australian average) this would be a savings of over $110 000-330 000 per year based on 10-30% dose reduction.

The negative aspects of changing include the pain patients will experience with injections and the potential for non-compliance if the erythropoietin is self-administered. Therefore, the Renal Unit at Sir Charles Gairdner Hospital has decided to convert all hemodialysis patients receiving IV ESA to SC administration in the belief that this will provide a considerable cost saving. Adjustments of doses will remain with the individual caring physicians, along the lines of usual clinical practice or a 'real-life' setting. We wish however to monitor the epoetin dose changes achieved in an Australian setting to ensure that dose reductions are achieved and that this does not occur as the expense of better anemia management. We plan to monitor this through the audit process.

Subjects and Methods

All conventional hemodialysis patients currently dialysing in the Sir Charles Gairdner Hospital (SCGH) Dialysis Programs will convert from intravenous to subcutaneous administration of ESA. Those currently on IV epoetin alfa will be converted to either SC epoetin alfa or SC epoetin beta. Those patients on IV darbepoetin alfa will convert to SC darbepoetin alfa. Conversion to SC epoetin formulations will be based upon a 80-100% dose conversion factor, to ensure patient Hb does not fall below 11.0 g/dL and to allow estimation of the conversion factor from IV to SC in an Australian clinical practice setting. There will be no dose reduction with SC darbepoetin alfa. The ESA will continue to be administered by the dialysis nurse with the initial dosing schedule being no more frequent than once per week. If patients move between dialysis units they will remain treated with their allocated ESA.

This study will follow standard clinical practice. As such, dose changes of ESA will be made by the patients' usual treating nephrologist according to their usual practice patterns. Intravenous iron protocols currently exists in all of these dialysis units and will continue. Anemia coordinators currently monitor hemoglobin and iron studies on all of these dialysis patients with the variables required being entered into a database. Routine unit-based quality monitoring will continue according to current practices.

ELIGIBILITY:
Inclusion Criteria:

* On haemodialysis at a Sir Charles Gairdner Hospital Unit

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil C Boudville, MBBS, Study Director — Sir Charles Gairdner Hospital
Locations (1):
- Sir Charles Gairdner Hospital, Perth, Western Australia, Australia